CLINICAL TRIAL: NCT04790994
Title: COVID-19 Prevalence in UNIVI Group Nursing Homes and Geriatric Healthcare Institutions: Epidemiological Study of Immunological Status With Rapid Serological Tests for Diagnostic Guidance
Brief Title: COVID-19 Prevalence in UNIVI Geriatric Institutions: Epidemiological Study of Immunological Status With Rapid Serological Tests
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Médical Porte Verte (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A01838-31
Record Dates: First submitted 2021-02-10; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-02

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To date, little information is available on the prevalence of Covid-19 and data are lacking on the proportion of patients, institutional residents and caregivers who have actually been exposed to SARS Cov-2.

With the NG Biotech rapid serological test, an individual's immunological status (presence of IgM and IgG antibodies) can be determined in 15 minutes on a finger-prick blood sample.

The proposed trial will be a noninterventional study of immunological status among the residents and caregivers of 26 nursing homes and 4 geriatric healthcare institutions belonging to the UNIVI Group who are representative of the institutional geriatric population in France. The NG Biotech rapid test will be carried out concomitantly with polymerase chain reaction (PCR) tests performed within the framework of a national screening campaign. Data on risk factors in staff members and on specific COVID 19 symptoms in residents will also be collected.

The study will terminate for residents and caregivers whose tests are both negative (absence of infection and no exposure to the virus). For residents and caregivers who have at least one positive test, follow-up visits will be scheduled in order to study the serology time course and the occurrence of reinfection (follow-up questionnaire).

DETAILED DESCRIPTION:
Type of study: multicentric prospective observational Study location: 26 nursing homes and 4 geriatric hospitals belonging to the UNIVI Group in France

Context:

At the end of the Covid-19 containment period in France, data published by Public Health France revealed that frail and dependent elderly people in nursing homes and geriatric healthcare institutions had paid a heavy tribute. As of May 4, 2020, the majority of reported Covid-19 cases (n=4,600; 63%) had occurred in nursing home residents and more than one-third (n=2,664; 37%) in patients in geriatric healthcare institutions. A total of 71,216 Covid-19 cases of which 33,948 (48%) were confirmed by reverse transferase polymerase chain reaction (RT-PCR) tests were reported to health authorities (Agence Régionale de Santé, ARS). Among reported cases, there were 12,726 deaths. Three-quarters of these deaths (9,501; 75%) occurred in geriatric institutions, the vast majority (99%) in nursing homes and 3,321 (25%) in hospitals. Reports of infection among staff members of these institutions reached 39,294 cases, of which 18,175 (46%) were confirmed by RT- PCR.

The confinement allowed a significant and continuous decrease in the number of Covid cases in French geriatric institutions since the beginning of April. The proportion of new cases observed among institutionalized geriatric residents has since fallen sharply, particularly in the most affected geographic regions. This is why deconfinement should be gradual and should be constantly reassessed on the basis of national and regional epidemiological data. Each nursing home should to take into account its own daily data showing the number of new diagnoses or suspected cases among residents and caregivers, keeping in mind the risk of transmission by visitors in the event of a recurrence of the epidemic.

In France, the deconfinement strategy began on April 20, 2020 in Île-de-France. Family visits under strict conditions were authorized in geriatric institutions. Currently, the modus operandi is accompanied by a PCR test campaign in order to have an inventory of the COVID status of all institutional residents and caregivers. Thus, any resident with a positive PCR test will be isolated until recovery and any caregiver with a positive PCR test will be quarantined.

For nursing home admissions, in accordance with ARS guidelines, a PCR test may be requested upon prescription from the institution's coordinating physician. Room confinement for newly admitted residents will be determined by the institution's geographical localization. Administrative districts are classified in two zones, red and green. For institutions in the red zone, room confinement with close medical supervision is compulsory for 14 days, corresponding to the viral incubation time. For institutions in the green zone, room confinement is not mandatory, but close medical surveillance is recommended.

What could NG Biotech rapid serological tests bring to the deconfinement strategy? These tests make it possible to determine an individual's immunological status (presence of IgM and IgG antibodies) in 15 minutes on a finger-prick blood sample. The test cannot be used in the acute phase of the disease, but makes it possible to confirm the serological status of an asymptomatic patient 15 days after the first clinical signs. Test sensitivity (ability to identify antibodies) is 100%. Serological testing does not answer the same question as PCR. PCR directly detects the presence of the virus, optimal in the first 7 days, it can remain positive for up to 3 weeks or even beyond. The serological test provides information on whether or not there is contact with the virus. If the serological test is positive in an asymptomatic patient, the patient is likely more than 15 days from symptom onset. It does not provide information on the risk of contagiousness. For nursing homes and geriatric healthcare institutions, use of serological testing, common law is applicable. The superior French health agency (Haute Autorité de Santé, HAS) specifies that these tests are indicated for epidemiological study or as a diagnostic catch-up tool (Place of rapid serotests in the strategy for the management of the COVID-19, HAS, May 14, 2020). The HAS recommendation specifies that rapid diagnostic tests must be performed by: - Professionals and staff who have previously received training in the use of COVID-19 rapid diagnostic tests - Doctors practicing in private practice - Doctors, medical biologists, midwives working in an institution or in a healthcare service (e.g. specialized screening structures) - Nurses or laboratory technicians working in an institution or in a healthcare service under the supervision of a doctor or a medical biologist - Midwives or nurses working in a prevention structure or an associative structure involved in health prevention - Community pharmacists - Employees or volunteers, non-healthcare professionals working in a prevention structure or an association structure, provided that they have previously received training in the use of rapid diagnostic tests.

To date, little information is available on the prevalence of Covid-19 and data are lacking on the proportion of patients, institutional residents and caregivers who have actually been exposed to SARS Cov-2. Likewise, in the scientific literature, there is uncertainty among people who have acquired immunity as to the persistence of neutralizing antibodies at 6 months and the risk of re-infection with COVID 19 after a primary infection. A major campaign of serological tests is in preparation in the geriatric institutions of the UNIVI Group. This study is based on this campaign using data collected in 26 nursing homes and 4 geriatric healthcare institutions. In total, around 2,000 residents, and 2,000 caregivers will be tested. The residents and caregivers of the tested institutions are representative of the institutionalized geriatric population in France. It is thus proposed to carry out a non-interventional study among residents and caregivers in nursing homes and in healthcare institutions belonging to the UNIVI Group. NG Biotech rapid tests will be performed concomitantly with PCR tests made within the framework of the national screening campaign.

ELIGIBILITY:
Inclusion Criteria:

* Residents of participating nursing home - who benefited from a rapid diagnostic orientation serological test for COVID-19 - having given their agreement
* All staff members (doctors, nurses, health executives, caregivers, physiotherapists, ASH, stretcher bearers, psychologists, dieteticians, administrative staff, secretaries, ...) - who benefited from a rapid diagnostic orientation serologic test for COVID-19 - having given their agreement

Exclusion Criteria:

* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 1145 residents and 1134 professionals in 26 nursing homes and 4 geriatric hospitals
Sampling Method: Probability Sample
Enrollment: 1145 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2021-04-16 (Estimated)

PRIMARY OUTCOMES:
Among asymptomatic residents and caregivers in French nursing homes and geriatric healthcare institutions belonging to the UNIVI Group: prevalence of covid 19 | three months
  positive RT-PCR test and/or (for residents) clinical diagnosis recorded in the medical file
Exposure to SARS Cov-2 Among asymptomatic residents and caregivers in French nursing homes and geriatric healthcare institutions belonging to the UNIVI Group | three months
  positive NG Biotech rapid serological test

SECONDARY OUTCOMES:
Recurrence of Covid-19 at 1, 3 and 6 months among residents and caregivers who had at least on positive test at inclusion (RT-PCR test or NB Biotech rapid serological test) | Time Frame: one, three and six months after inclusion]
  RT-PCR in favor of Covid-19 recurrence and/or positive results of an NG Biotech rapid serological test.
Risk factors for Covid-19 infection in caregivers | three months
  analysis of the questionnaire items: age; sex; occupation; type of housing; family composition; means of transportation; contact with an infected person
Covid-19 symptoms among residents | three months
  analysis of symptoms reported on the questionnaire
Prevalence of Covid-19 at 3 months | three months
  positive test (RT-PCR or NB Biotech rapid serological test) and/or (for residents) suspected or definitive diagnosis of Covid-19 recorded in the medical file.

CONTACTS AND LOCATIONS:
Locations (1):
- CentreMédicalPorteVerte, Versailles, France